CLINICAL TRIAL: NCT03910569
Title: Smidt Heart Institute Takotsubo Registry
Brief Title: The Cedars-Sinai Smidt Heart Institute Takotsubo Registry & Proteomic Study
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director of Women's Heart Center, Cedars-Sinai Medical Center
Other Study IDs: 53569
Record Dates: First submitted 2019-03-06; First posted 2019-04-10 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Takotsubo Cardiomyopathy
Keywords: Takotsubo
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples Without DNA — The blood samples will undergo proteomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Cedars-Sinai SHI Takotsubo Registry and Proteomic Study is an observational registry that will collect retrospective and prospective demographic, clinical, hemodynamic, laboratory and other diagnostic parameters, therapy and outcome data from individuals who meet the inclusion/exclusion criteria of Takotsubo Registry protocol. Subjects will also be invited to provide a blood sample utilizing a Mitra kit sent to their homes. Researchers from the Barbra Streisand Women's Heart Center will analyze Registry data to identify Takotsubo phenotypes, improve diagnostic capabilities, better predict recurrence rates, and develop targeted Takotsubo treatments.

DETAILED DESCRIPTION:
Registry outreach will begin with an informational and inspirational website and will utilize social media and patient-driven activism through Facebook, blogs and Twitter modalities that have demonstrated efficiencies in other patient-centered research efforts. Subjects will upload specific clinical materials into Cedar-Sinai's web-enabled cloud storage and which will be screened by trained Smidt Heart Institute physicians. The Registry utilizes on-line, e-consent and enrollment connected to a REDCap database that will allow efficient data input for analysis. All potential subjects who have been diagnosed with Takotsubo or have been informed by their physician that they meet diagnosis criteria, will need to provide information for review that includes: hospitalization records, from the time of Takotsubo event, with laboratory data (particularly -- troponin level), ECG and CTA. Registrants will be asked to respond to annual update surveys.

The goal is to accurately understand the prevalence, recurrence and prospective status of the Takotsubo, to determine which individuals are at risk of reoccurrence or subsequent adverse event and to determine potential treatment targets to develop therapeutic strategies

Primary:

* To establish a large USA-based database for patients with Takotsubo with a convenient and easy to use on-line patient-advocate registry using digital media marketing, Box cloud data access and storage, accurate case adjudication, and automated follow-up.
* Participants will also be offered the option of participating in the Takotsubo Proteomic Registry by providing remote ambulatory Mitra blood samples.

Secondary:

• To establish a clinical trial platform for patient-centered point-of-care trials to improve diagnostics, clinical care and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have received a diagnosis of Takotsubo from their physician and consent to enroll
* Submit full medical records needed for Takotsubo adjudication

Exclusion Criteria:

* Younger than 18 years
* Unable to provide informed consent
* Unable to provide the necessary documentation needed for screening purposes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The registry will be open to all subjects who have experienced a diagnosed Takotsubo syndrome episode or have been informed by their treating physicians that they have the syndrome.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Prevalence of the Takotsubo | Baseline, Annual follow-up up to 30years
  Prevalence of the Takotsubo will be measured annually. Change from baseline will be assessed.
Number of participants with Recurrence the Takotsubo | Baseline, Annual follow-up up to 30years
  Recurrence the Takotsubo will be measured annually. Change from baseline will be assessed.
Annual update surveys will collect data on patient's prospective health status following Takotsubo event | Baseline, Annual follow-up up to 30years
  Prospective statusof the Takotsubo will be measured annually. Change from baseline will be assessed.
Risk factors affecting which patients, having had one Takotsubo event, will more likely experience a Takotsubo reoccurrence or related subsequent adverse event | Baseline, Annual follow-up up to 30years
  Risk factors for reoccurrence or subsequent adverse event will be collected annually.

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, FACC, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marano P, Maughan J, Obrutu O, Lauzon M, Tjoe B, Herscovici R, Moy P, Rojas N, Shufelt C, Rutledge T, Wei J, Bairey Merz CN. Evaluation of Recurrent Takotsubo Syndrome. JACC Adv. 2024 Sep 17;3(10):101247. doi: 10.1016/j.jacadv.2024.101247. eCollection 2024 Oct. PMID 39324115